CLINICAL TRIAL: NCT00342186
Title: Human Genes Involved in Susceptibility or Resistance to Hepatitis B Virus
Brief Title: Genes Involved in Resistance or Susceptibility to Hepatitis B Virus
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902323; 02-C-N323; NCT00565825 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hepatitis, Viral, Human
Keywords: China; Cancer; Hepatitis B; Genetics; Liver Disease; HBV
MeSH Terms: conditions — Hepatitis, Viral, Human; Neoplasms; Hepatitis B; Liver Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

SUMMARY:
This study, conducted by the Beijing University First Hospital of China and the National Cancer (NCI), will try to identify genes associated with either susceptibility or resistance to chronic infection by the hepatitis B virus (HBV). Some people recover from HBV infection; others become chronically infected and may go on to develop severe liver disease such as cirrhosis or liver cancer. About 350 million people worldwide have chronic HBV infection. Of 120 million infected Chinese, 90 percent of children infected at less than 5 years of age and 10 percent of infected adults develop persistent infection.

HBV-infected and non-infected healthy persons of Han ethnicity born before 1963 may be eligible for this study. Offspring of infected candidates (born in any year) may also be enrolled. Infected adults must have at least one infected parent or sibling. Persons who resided in Fusui County of Guangxi Zhuang Autonomous Region or in the Qidong district of Jiangsu Province for at least 6 months before 1986 may not participate.

All participants (except offspring of the study subjects) will fill out a health questionnaire (providing information about eating, drinking, and smoking habits and a personal and family health history) and will donate no more than 20 milliliters of blood. The blood will be tested for antibodies, antigens, and other substances that may indicate infection with hepatitis viruses. Some of the blood will be sent to the NCI for DNA analysis to identify genetic factors that may influence clearance of the hepatitis virus after infection or progression to liver diseases associated with HBV infection. Infected patients who have had a liver biopsy in the past will be asked permission to examine tissue from the biopsy and to review laboratory results of any tests done for diagnostic and treatment purposes.

When the study is completed, specimens sent to the NCI will have identifiers linking the material to the donor removed. The anonymous samples may then be used for other genetic studies. Specimens remaining in China will continue to have identifiers linked to them and may be used for future studies designed to identify who is at greatest risk of developing serious liver diseases. Participants who do not want their blood used for future studies may request that the samples be destroyed.

Because children inherit one-half of their DNA from each parent, DNA samples from HBV infected study participants may provide additional information about the parent s DNA structure. Offspring who participate in this study will provide a DNA sample. The sample is obtained by swishing a mouthwash in the mouth for 30 seconds and then spitting the mouth wash into a cup. The DNA is then isolated from the mouth cells.

DETAILED DESCRIPTION:
Persistent hepatitis B viral (HBV) infection is a significant public health problem because of the occurence of chronic liver disease, cirrhosis, and hepatocarcinoma (HCC) [1-3]. Roughly one-third of the world population has been infected with HBV and there are about 350 million (5-6%) persistent carriers. HBV causes 80% of all liver cancer and is the second most important carcinogen, after smoking tobacco. There is an approximate 90% risk of becoming a persistent carrier following perinatal infection in infants born to e antigen positive carrier mothers and 30% risk in pre-school children. Only 5-10% of adults become persistent carriers following infection. Like HIV, HBV is transmitted by contaminated blood through transfusion or intravenous drug use and by high-risk sexual behavior.

The purpose of this investigation is to study how different outcomes of hepatitis B exposure and infection are affected by host genetic factors in the Chinese population, where more than 120 million individuals are infected with HBV. Of people persistently infected with HBV, 10-30% will develop liver cirrhosis (LC) and hepatocellular carcinoma (HCC). These highly variable outcomes in both clearance rates and disease outcomes in persistently infected individuals cannot be fully explained by differences in viral or environmental factors. Thus, differences in host genetic factors may affect hepatitis B natural history.

Blood will be collected from volunteers in China. Healthy donors unexposed to HBV or HCV, individuals who have cleared HBV, and asymptomatic carriers of HBV will be identified by the Peking University hospitals and blood bank. HBV infected individuals with chronic hepatitis, cirrhosis or HCC will be identified by the Peking University hospital hepatitis clinics. Targeted individuals will be asked to participate by letter or a telephone interview by trained hospital staff. A database of clinical and family information will be created from a questionnaire completed by hospital staff. A database of clinical and family information will be created from a questionnaire completed by hospital staff interviewers. Blood will be separated into plasma and peripheral blood mononuclear cells (PBMCs) and cryopreserved in China. Serum will be tested in China for hepatitis viral markers, HBV genotypes, and HBV viral load. Two vials of PBMC will be transferred to the LGD, NCI-USA, for mRNA expression assays and host genetic analysis. Lymphoblastoid cell lines will be established by the LGD-NCI as a source of renewable DNA. RNA will be extracted from PBMCs for determination of mRNA expression by the microarray method. Results of mRNA expression assays and literature searches will be used to identify candidate genes. DNA extracted from cell lines will be genotyped for single nucleotide polymorphisms (SNPs) in candidate genes and DNA markers, including HLA, cytokines, chomokines, and their receptors, and putative HBV cell entry targets by DNA genotyping methods. SNPs in candidate genes will be identified using public and private SNP databases and SNP discovery methods. SNPs will be genotyped study participants and analyzed to detect associations between polymorphisms and phenotypes obtained from clinical and laboratory testing. If a genetic marker associated with the development of a disease phenotype is found, there are potential applications in diagnostics and therapy. The identification of allelic polymorphisms in genes involved in the pathway from chronic viral infection to LC and ultimately HCC would provide insight into the carcinogenic process.

ELIGIBILITY:
* INCLUSION CRITERIA:

A Group - HBV Clearance:

1. HBsAg negative and anti-HBs and anti-HBc positive or anti-HBs positive and no HB Vaccination history.
2. No systemic diseases.

B Group - Asymptomatic persistent infection:

1. HBsAg, anti-HBc positive for at least 6 months.
2. At least one parent or sibling HBsAG positive .
3. ALT and AST have been in normal range (less than 45 IU/L) at least 5 years
4. No clinical symptoms of hepatitis.
5. No clinical liver cirrhosis.

C Group - Chronic Hepatitis B:

1. HBsAg, anti-HBc positive for more than 6 months.
2. At least one parent or sibling HBsAg positive.
3. ALT and/or AST were greater than or equal to 60 IU/L or greater than 2 times upper limit of normal.
4. No clinical liver cirrhosis.
5. No other systemic diseases.

D Group - Decompensated liver cirrhosis:

1. HBsAg and anti-HBc positive.
2. At least one parent or sibling HbsAg positive.
3. Decompensated liver cirrhosis (gastroesophageal varication, ascites or edema)

E Group - Primary hepatocellular carcinoma:

1. HbsAg or anti-HBc positive.
2. At least one parent or sibling HBsAg positive.
3. HCC confirmed by liver biopsy or by both AFP an ultrasound, CT or MRI.

F Group - Normal Donor Group:

1. HbsAg negative and anti-HBc and anti-HBs negative
2. ALT and AST are in normal range (less than 45 IU/L)
3. No systemic diseases.

Offspring of cases (for haplotype determinations):

1. Natural child of cases.
2. Age 8 or older.

EXCLUSION CRITERIA:

B thru E Groups:

1. Persons born in 1963 or later.
2. Persons not of Han ethnicity.
3. Persons with no first-order relative (parent or sibling) with HBV infection.
4. Persons who resided in Fusui County of Guangzi Zhuang Autonomous Region or in the Qidong district of Jiangsu Province for at least 6 months prior to 1986.
5. anti-HCV, HCV RNA, anti-HDV, and/or HDAg.
6. Current infection with HAV or HEV (indicated by antibodies and abnormal liver function).
7. Persons meeting the inclusion criteria but who are unwilling or unable to give informed consent.

A & F Groups - HBV Clearance & Normal Donors:

1. Persons born in 1963 or later.
2. Persons not of Han ethnicity.
3. Persons who resided in Fusui County of Guangxi Zhuang Autonomous Region or in the Qidong district of Jiangsu Province for at least 6 months prior to 1986.
4. Anti-HCV, HCV RNA, anti-HDV and/or HGAg positive.
5. Current infection with HAV or HEV (indicated by antibodies and abnormal liver function).
6. Persons meeting the inclusion criteria but who are unwilling or unable to give informed consent.

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthy donors and those infected with HBV
Sampling Method: Non-Probability Sample
Enrollment: 2303 (Actual)
Dates: Start 2002-09-27 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Collection of 3400 samples | Annual
  genotyping study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W McVicar, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Peking University First Hospital, Beijing, China

REFERENCES:
- [Background] Risch N, Merikangas K. The future of genetic studies of complex human diseases. Science. 1996 Sep 13;273(5281):1516-7. doi: 10.1126/science.273.5281.1516. No abstract available. PMID 8801636
- [Background] O'Brien SJ, Nelson GW, Winkler CA, Smith MW. Polygenic and multifactorial disease gene association in man: Lessons from AIDS. Annu Rev Genet. 2000;34:563-591. doi: 10.1146/annurev.genet.34.1.563. PMID 11092839
- [Background] Chisari FV. Cytotoxic T cells and viral hepatitis. J Clin Invest. 1997 Apr 1;99(7):1472-7. doi: 10.1172/JCI119308. No abstract available. PMID 9119989